CLINICAL TRIAL: NCT03320759
Title: Enhancing Recovery in Non-Traumatic Spinal Cord Injury: Implementation of an Integrated Program for the Assessment of Rehabilitation Therapies
Brief Title: Enhancing Recovery in Non-Traumatic Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 108706
Record Dates: First submitted 2017-09-27; First posted 2017-10-25 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Compression; Spinal Cord Injuries; Cervical Spondylosis; Myelopathy Cervical
MeSH Terms: conditions — Spinal Cord Compression; Spinal Cord Injuries; Spondylosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No rehabilitation (No Intervention)
- Rehabilitation (Experimental)
  Interventions: Behavioral: Occupational therapy rehabilitation

INTERVENTIONS:
Behavioral: Occupational therapy rehabilitation — Participants in the experimental arm will receive occupational therapy that is individualized to each participant's needs from week 4 post-decompression surgery until week 12.
  Arms: Rehabilitation

SUMMARY:
The investigators have spent the last decade uncovering unique metabolic and functional abnormalities in the brains of patients with spinal cord compression. Degenerative spinal cord compression represents a unique model of reversible spinal cord injury. In the investigator's previous work, they have demonstrated that cortical reorganization and recruitment is associated with metabolic changes in the brains of patients recovering from spinal cord compression and is correlated with recovery and improved neurological scores.

The goal of this study is to combine a rigorous platform of clinical care that includes preoperative evaluation, surgery, and rehabilitation, with state of the art imaging techniques to demonstrate how rehabilitative therapy can increase brain plasticity and recovery of neurological function in patients with spinal cord injury. Neurological function will be carefully evaluated in two groups of patients, those receiving rehabilitation and those not receiving rehabilitation after spine surgery, and will be correlated with the results of advanced imaging.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* have a history of progressive neurological deficits <24 months
* eligible for MRI scanning

Exclusion Criteria:

* having any other neurological disorder or systemic disease that can impair neurological function
* not fluent in reading and speaking English
* being claustrophobic
* unable to follow simple task instructions and maintain standardized movements
* being unable to return for all follow-up imaging and rehabilitation sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in levels of N-acetylaspartate (NAA) in the motor cortex | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)
  It is expected that the group of patients receiving rehabilitation will experience less decline in NAA concentrations as compared to the second group of patients not receiving rehabilitation.
Changes to volume of activation in motor and supplementary motor cortices | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)
  Volume of activation is measured by calculating the voxel number within our selected cortical regions, the motor cortex and supplementary motor cortex, using functional magnetic resonance imaging (fMRI). Changes in these numbers demonstrate volume of cortical activation changes in these regions. Following rehabilitation, the investigators expect that the volume of cortical activation of patients, expressed as voxel number, will change between time points compared with changes observed in the control group.
Changes in Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) scores | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)
  Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) is an indicator of dorsal and palmar sensation, strength (by myotome) and prehension (grasping). GRASSP is a standardized measure to assess hand function in ways that are meaningful in the context of a patient's overall ability to complete activities of daily living.
Changes to intensity of cortical activation in motor and supplementary motor cortices | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)
  Intensity of cortical activation is expressed as signal intensity in beta weights. Following rehabilitation, the investigators expect that the intensity of cortical activation in participants in the intervention group will change between time-points compared with changes observed in the control group.

SECONDARY OUTCOMES:
RAND Short form (SF)-36 Health Survey Questionnaire | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)]
  General health status self-administered evaluation tool. Better scores in the intervention group are expected. Composite score will be reported. The range for this score is from 0 to 100, with 100 indicating the best general health status possible. Subscale scores also range from 0-100 and are simply an average of the scores for each of their relevant questions. Subscales are combined into a composite score by averaging results of all subscales, which is the methodology specified by the creators of the scale (RAND).
Modified Japanese Orthopaedic Association (mJOA) scale | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)
  A clinical tool used to evaluate impairment due to cervical spondylotic myelopathy, including loss of sensation, motor abilities in limbs, and bowel and bladder control. The lowest possible score is a 0 and the highest, 18. Higher numbers indicate better functioning. Item scores are simply summed to arrive at the composite score.
Myelopathy Disability Index (MDI) | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)
  This self-administered questionnaire is used to measure the degree to which myelopathy has affected the participant's ability to perform activities of daily living. Raw scores will be calculated for each participant and may range from 0 to 30. To arrive at the participant's raw score, item scores are simply summed. The final scores used for analysis will be the participant's score expressed as a percentage. Higher scores indicate greater impairment.
American Spinal Injury Association (ASIA) Impairment Scale | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)
  A clinical assessment tool used to classify motor and sensory impairment in persons with myelopathy. Subscales to be reported include the right and left motor scores (range=0-50 for both) and the right and left sensory scores (range=0-60 for both). Higher scores indicate less impairment.
Strength as tested with hand dynamometer | Measured and reported for all follow-ups throughout study (i.e. pre-operatively, 4 weeks, 6 weeks, 6 months)
  A device used to measure grip strength.

CONTACTS AND LOCATIONS:
Locations (1):
- LHSC - University Hospital, London, Ontario, Canada